CLINICAL TRIAL: NCT06788990
Title: A Multicenter, Randomized, Double-blind, Phase 2/3 Study of Ficerafusp Alfa (BCA101) or Placebo in Combination With Pembrolizumab for First-Line Treatment of PD-L1-positive, Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: FORTIFI-HN01: A Study of Ficerafusp Alfa (BCA101) or Placebo in Combination With Pembrolizumab in First-Line PD-L1-pos, R or M HNSCC
Acronym: FORTIFI-HN01
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bicara Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCA101X301; 2024-519654-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-10; First posted 2025-01-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: Phase 2/3; Ficerafusp alfa; BCA101; Recurrent Head and Neck Squamous Cell Carcinoma (R HNSCC); Metastatic Head and Neck Squamous Cell Carcinoma (M HNSCC); Pembrolizumab; EGFR; TGF-beta
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Camurati-Engelmann Syndrome | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 2 Arm A (Experimental): ficerafusp alfa 1500 mg QW + pembrolizumab 200 mg every 3 weeks (Q3W)
  Interventions: Drug: Ficerafusp alfa; Drug: Pembrolizumab (KEYTRUDA®)
- Phase 2 Arm B (Experimental): ficerafusp alfa 750 mg QW + pembrolizumab 200 mg Q3W
  Interventions: Drug: Ficerafusp alfa; Drug: Pembrolizumab (KEYTRUDA®)
- Phase 2 Arm C (Placebo Comparator): placebo QW + pembrolizumab 200 mg Q3W
  Interventions: Drug: Pembrolizumab (KEYTRUDA®); Drug: Placebo
- Phase 3 OBD Arm (Experimental): ficerafusp alfa OBD + pembrolizumab 200 mg Q3W
  Interventions: Drug: Ficerafusp alfa; Drug: Pembrolizumab (KEYTRUDA®)
- Phase 3 Arm C (Placebo Comparator): placebo QW + pembrolizumab 200 mg Q3W
  Interventions: Drug: Pembrolizumab (KEYTRUDA®); Drug: Placebo

INTERVENTIONS:
Drug: Ficerafusp alfa — Investigational
  Arms: Phase 2 Arm A; Phase 2 Arm B; Phase 3 OBD Arm
Drug: Pembrolizumab (KEYTRUDA®) — Immunotherapy agent used in combination with investigational agent
Drug: Placebo — Placebo Control
  Arms: Phase 2 Arm C; Phase 3 Arm C

SUMMARY:
Ficerafusp alfa is directed against two targets, Epidermal Growth Factor Receptor (EGFR) and Transforming Growth Factor beta (TGF-β).

This study intends to evaluate the safety and efficacy of ficerafusp alfa in combination with pembrolizumab versus placebo with pembrolizumab in 1L PD-L1-positive, recurrent or metastatic Head and Neck Squamous Cell Carcinoma (HNSCC).

DETAILED DESCRIPTION:
The mechanism of action of ficerafusp alfa involves dual targeting of two cancer targets, EGFR and TGF-β, which are known to drive solid tumor growth and metastasis.

Phase 2 of the study will identify an optimal biologic dose (OBD) supported by the safety, tolerability, PK, PD, and efficacy data of ficerafusp alfa. In this part, eligible subjects will be randomized to one of three treatment arms at a 1:1:1 ratio:

* Arm A: ficerafusp alfa 1500 mg once weekly (QW) + pembrolizumab 200 mg every three weeks (Q3W).
* Arm B: ficerafusp alfa 750 mg QW + pembrolizumab 200 mg Q3W.
* Arm C (control): placebo QW + pembrolizumab 200 mg Q3W.

The primary objective for the phase 3 portion is to compare the efficacy in subjects treated with ficerafusp alfa at the selected OBD in combination with pembrolizumab versus placebo with pembrolizumab. Eligible subjects will be randomized 2:1 in the treatment versus control arm during the phase 3 portion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years on the day the Informed Consent Form is signed.
* Histologically or cytologically confirmed R or M HNSCC. Eligible primary tumor locations are oral cavity, hypopharynx, larynx or oropharynx (with documented HPV-negative disease if presenting with OPSCC). Note: primary tumor location of paranasal sinuses and nasopharynx, any histology are excluded.
* No prior systemic therapy administered in the R or M setting; and completed systemic therapy >6 months prior if given as part of multimodal treatment for locoregionally advanced disease in the adjuvant or definitive setting.
* Archival tumor tissue or willing to undergo pretreatment biopsy at Screening if archival tissue is insufficient or unavailable.
* PD-L1 CPS ≥1 (by PD-L1 IHC 22C3 pharmDx assay).
* Measurable disease based on RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function, as defined in the protocol.

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent.
* Prior treatment with anti-TGFβ therapy.
* Prior therapy with an anti-EGFR antibody (exception: radio sensitizing agents and multimodal treatment for locoregionally advanced disease).
* Prior history of Grade ≥2 intolerance or hypersensitivity reaction to anti-EGFR therapy or other murine proteins.
* Prior therapy with an immune checkpoint inhibitor completed within 6 months prior to study treatment initiation.
* Progressive disease <6 months from completion of curative intent systemic therapy for locoregionally advanced HNSCC.
* Life expectancy less than 3 months.
* Known active central nervous system metastases, history of spinal cord compression from tumor involvement, a history of carcinomatous meningitis, or leptomeningeal disease are excluded.
* Current active major bleeding, or a recent major bleeding episode within 4 weeks prior to enrollment.
* Subject participated in another clinical study or received treatment with another investigational drug must wait at least 5 half-lives of the treatment received or 4 weeks (whichever is shorter) following prior therapy.
* Active autoimmune disease requiring systemic treatment in the past 2 years.
* Subjects with chronic hepatitis B virus (HBV) infection with active disease who meet the criteria for anti-HBV therapy and are not on a suppressive antiviral therapy prior to initiation of study treatment.
* Subjects with a known history of hepatitis C virus (HCV) who have not completed curative antiviral treatment or have an HCV viral load above the limit of quantification at Screening.
* Known history of human immunodeficiency virus (HIV).
* Receipt of any organ transplantation, including autologous and allogeneic stem cell transplantation, with the exception of transplants that do not require immunosuppression.
* Known to be diagnosed and/or treated for any other additional malignancy within 2 years prior to randomization with the exception of the following: curatively treated basal cell carcinoma or squamous cell carcinoma of the skin, and curatively resected in situ cervical cancer, and curatively resected in situ breast cancer, and low-risk early stage prostate cancer.
* Any condition requiring systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication within 7 days prior to the first dose of study treatment, except for topical, intranasal, intrabronchial, or ocular steroids.
* Use of a live or live attenuated vaccine within 4 weeks prior to Screening.

Other Inclusion/Exclusion criteria may apply as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Phase 2 - Incidence and severity of TEAEs, treatment-treatment emergent SAEs TEAEs leading to dose interruption, dose reduction, or permanent discontinuation. | Up to 30 days post end of treatment for TEAEs (90 days for SAEs).
  To assess safety and tolerability of ficerafusp alfa with pembrolizumab.
Phase 2 - Objective Response Rate (ORR) per RECIST 1.1 by blinded independent central review (BICR) | Approximately 1 year.
  ORR is defined as the proportion of subjects in the DDS who have a confirmed CR or PR per RECIST 1.1. by BICR.
Phase 3 - Objective Response Rate (ORR) per RECIST 1.1 by BICR. | Approximately 2 years.
  ORR is defined as the proportion of subjects in the DDS who have a confirmed CR or PR per RECIST 1.1. by BICR.
Phase 3 - Overall Survival (OS) | Approximately 3 years.
  OS: Defined as the time from the randomization to death due to any cause.

SECONDARY OUTCOMES:
Phase 2 - Duration of Response (DOR) per RECIST 1.1 by BICR. | Approximately 1 year.
  DOR: For subjects who demonstrated CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death, whichever occurs first, per RECIST 1.1 by BICR.
Phase 3 - Incidence and severity of TEAEs, treatment-treatment emergent SAEs TEAEs leading to dose interruption, dose reduction, or permanent discontinuation. | Up to 30 days post end of treatment for TEAEs (90 days for SAEs).
  To assess safety and tolerability of ficerafusp alfa with pembrolizumab.
Phase 3 - Progression-free survival (PFS) per RECIST 1.1 by BICR. | Approximately 3 years.
  PFS: Defined as the time from randomization to the first documented PD per RECIST 1.1 as determined by BICR or death due to any cause, whichever occurs first.
Phase 3 - Objective Response Rate (ORR) per RECIST 1.1 by BICR. | Approximately 3 years.
  ORR: Defined as confirmed CR + PR per RECIST 1.1 by BICR. (FAS).
Phase 3 - Duration of Response (DOR) per RECIST 1.1 by BICR. | Approximately 3 years.
  DOR: For subjects who demonstrated CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death, whichever occurs first per RECIST 1.1 by BICR.
Phase 3 - Clinical Benefit Rate (CBR) per RECIST 1.1 by BICR. | Approximately 3 years.
  Clinical Benefit Rate: For subject who demonstrated CR + PR + SD>6 months per RECIST 1.1 by BICR.
Phase 3 - ORR, per RECIST 1.1 by investigator's assessment. | Approximately 3 years.
  ORR, per RECIST 1.1 as determined by investigator's assessment.
Phase 3 - DOR, per RECIST 1.1 by investigator's assessment. | Approximately 3 years.
  DOR, per RECIST 1.1 as determined by investigator's assessment.
Phase 3 - PFS, per RECIST 1.1 by investigator's assessment. | Approximately 3 years.
  PFS, per RECIST 1.1 as determined by investigator's assessment.
Phase 3 - 14. Time to deterioration (TTD) in global health status measured by the EORTC QLQ C30 items for global health status and quality of life scale (item 29/30) | Approximately 3 years.
  To evaluate TTD in global health status/quality of life in subjects treated with ficerafusp alfa in combination with pembrolizumab versus placebo plus pembrolizumab.
  TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline in QoL using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30 Item 30) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher value indicates a better level of function.
Phase 3 - Time to deterioration (TTD) in pain measured by the EORTC HN 35 (items 31-34) pain domain. | Approximately 3 years.
  To evaluate TTD in pain in subjects treated with ficerafusp alfa in combination with pembrolizumab versus placebo plus pembrolizumab.
  TTD defined as the time from first dose (baseline) to change in pain score by 10-point from baseline, using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core Head and Neck Module (EORTC HN35). A higher score indicates a higher level of symptom burden.

CONTACTS AND LOCATIONS:
Locations (111):
- United States (49):
  - Site # 0137, Birmingham, Alabama
  - Site #0147, Phoenix, Arizona
  - Site #0107, La Jolla, California
  - Site #0106, Los Angeles, California
  - Site#0144, Sacramento, California
  - Site #0130, San Francisco, California
  - Site #0150, Stanford, California
  - Site #0122, Aurora, Colorado
  - Site #0124, Aurora, Colorado
  - Site#0121, Aurora, Colorado
  - Site#0127, Newark, Delaware
  - Site #0148, Jacksonville, Florida
  - Site #0136, Palm Bay, Florida
  - Site #0105, Tampa, Florida
  - Site #0133, Chicago, Illinois
  - Site#0140, Iowa City, Iowa
  - Site #0149, Westwood, Kansas
  - Site#0109, Lexington, Kentucky
  - Site#0111, Louisville, Kentucky
  - Site#0115, Louisville, Kentucky
  - Site #0112, Baltimore, Maryland
  - Site #0131, Boston, Massachusetts
  - Site#0101, Boston, Massachusetts
  - Site #0156, Maplewood, Minnesota
  - Site #0146, Rochester, Minnesota
  - Site #0114, St Louis, Missouri
  - Site #0119, Hackensack, New Jersey
  - Site #0155, New York, New York
  - Site#0142, New York, New York
  - Site#0118, Durham, North Carolina
  - Site#0154, Canton, Ohio
  - Site#0117, Cincinnati, Ohio
  - Site #0151, Cleveland, Ohio
  - Site #0108, Cleveland, Ohio
  - Site #0113, Portland, Oregon
  - Site #0103, Pittsburgh, Pennsylvania
  - Site #0123, Pittsburgh, Pennsylvania
  - Site #0132, Providence, Rhode Island
  - Site#0104, Charleston, South Carolina
  - Site#0126, Nashville, Tennessee
  - Site #0116, Nashville, Tennessee
  - Site#0102, Houston, Texas
  - Site #0152, Waco, Texas
  - Site#0134, Charlottesville, Virginia
  - Site #0129, Richmond, Virginia
  - Site #0138, Richmond, Virginia
  - Site #0125, Seattle, Washington
  - Site#0120, Vancouver, Washington
  - Site #0141, Madison, Wisconsin
- Australia (8):
  - Site#0302, Camperdown, New South Wales
  - Site #0306, Kingswood, New South Wales
  - Site#0304, Waratah, New South Wales
  - Site #0305, Southport, Queensland
  - Site#0307, Tugun, Queensland
  - Site #0303, Heidelberg, Victoria
  - Site#0301, North Melbourne, Victoria
  - Site#0308, Murdoch, Western Australia
- Austria (2):
  - Site #1602, Salzburg
  - Site #1601, Vienna
- Belgium (5):
  - Site #1007, Bruges
  - Site #1005, Mons
  - Site #1002, Namur
  - Site #1003, Namur
  - Site #1001, Sint-Niklaas
- Canada (2):
  - Site #0202, Vancouver, British Columbia
  - Site #0203, Montreal, Quebec
- France (5):
  - Site #0809, Amiens
  - Site #0807, Saint-Grégoire
  - Site #0808, Strasbourg
  - Site #0806, Vandœuvre-lès-Nancy
  - Site #0801, Villejuif
- Germany (2):
  - Site #0710, Aachen
  - Site #0706, Düsseldorf
- Site #0602, Dublin, Ireland
- Italy (6):
  - Site #0911, Florence
  - Site #0907, Milan
  - Site #0915, Napoli
  - Site #0908, Palermo
  - Site #0918, Rome
  - Site #0906, Rome
- New Zealand (2):
  - Site #0401, Christchurch
  - Site#0402, Rotorua
- Poland (5):
  - Site #1401, Gdansk
  - Site #1403, Katowice
  - Site #1407, Konin
  - Site #1404, Krakow
  - Site #1406, Warsaw
- Portugal (7):
  - Site #1506, Braga
  - Site #1503, Coimbra
  - Site #1508, Lisbon
  - Site #1501, Portimão
  - Site #1505, Porto
  - Site #1507, Porto
  - Site #1502, Senhora da Hora
- Spain (8):
  - Site #1301, Barcelona
  - Site #1305, Barcelona
  - Site #1304, Barcelona
  - Site #1310, Madrid
  - Site #1303, Madrid
  - Site #1306, Pamplona
  - Site #1309, Santander
  - Site #1307, Valencia
- United Kingdom (9):
  - Site #0504, Aberdeen
  - Site #0513, Cambridge
  - Site #0507, Liverpool
  - Site #0505, London
  - Site #0502, London
  - Site #0508, Manchester
  - Site #0503, Nottingham
  - Site #0515, Oxford
  - Site # 0501, Sutton